CLINICAL TRIAL: NCT02878928
Title: A Prospective, Multi-Center, Randomized Clinical Study to Evaluate the Clinical Impact of Pharmacogenetic-Guided Treatment for Depression & Anxiety
Brief Title: Clinical Study Evaluating Effects of Pharmacogenetic-guided vs Standard-of-Care Treatment on Depression and/or Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AltheaDx (Industry)
Collaborators: Innovis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CLP-0009
Record Dates: First submitted 2016-07-14; First posted 2016-08-25 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Depression; Anxiety
Keywords: Pharmacogenetic testing; PGx; Depression; Neuropsychiatric diseases; IDgenetix; AltheaDx
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDgenetix Neuropsychiatric Test Panel Intervention (Experimental): Medical providers for IDgenetix Neuropsychiatric Test Panel-guided group will make treatment recommendations based on test results. Patient outcomes will be measured throughout the duration of the study.
  Interventions: Genetic: IDgenetix Neuropsychiatric Test Panel
- Control Group (No Intervention): Medical providers for the Control Group will not receive IDgenetix Neuropsychiatric Test Panel results and will make treatment recommendations as usual. Patient outcomes will be measured throughout the duration of the study.

INTERVENTIONS:
Genetic: IDgenetix Neuropsychiatric Test Panel — The IDgenetix Neuropsychiatric Test Panel is used to make recommendations on the medication therapy that might be impacted by the genetic background of the patient.
  Other Names: PGx Testing
  Arms: IDgenetix Neuropsychiatric Test Panel Intervention

SUMMARY:
A prospective, multi-center, randomized, subject and outcome evaluator blind , parallel-group study evaluating the effect of pharmacogenetic-guided versus standard of care treatment for subjects diagnosed with depression and/or anxiety disorders.

DETAILED DESCRIPTION:
A substantial number of patients taking anti-depressant and anti-anxiety medications suffer from either a lack of benefit from drug therapy or severe side effects. Clinical features often fail to predict the drug response and tolerability of a patient to a prescription medication. Genetics can help guide therapeutic decisions for patients exhibiting neuropsychiatric disorders and potentially improve patient outcomes by maximizing drug efficacy and minimizing the risk of adverse events. Genetics and drug interactions can alter both the pharmacokinetics and pharmacodynamics of a multitude of drug compounds and in turn influence both the safety and efficacy of selected therapeutic regimens.

This study is designed to evaluate the clinical impact of pharmacogenetic (PGx)-directed treatment. Pharmacogenetic-guided therapy selection using the IDgenetix Neuropsychiatric Test Panel can enhance patient response and tolerability by facilitating the selection of the most appropriate medication at the most effective dose in the shortest possible time.

In this prospective, multi-center, randomized, subject and outcome evaluator blind, parallel-group study patients presenting to the clinical site with evidence of depression and/or anxiety as determined by a qualified clinician will be invited to participate. Study participants will be randomized to one of two groups with respect to the IDgenetix Neuropsychiatric Test Panel result: group with testing results revealed to the medical provider prior to treatment selection (Experimental Group) or group without testing results prior to treatment selection (Control Group). Participant outcomes will be measured at baseline and throughout the 3-month duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Subjects diagnosed with depression and/or anxiety as per the DSM-V criteria or standard of care site procedures and meeting at least one of the following:

  * Diagnosed with depression and/or anxiety either new to treatment or currently taking medications for less than 6 weeks.
  * Inadequately controlled with medications defined as inadequate efficacy after 6 weeks of a psychotropic treatment or have discontinued psychotropic treatment due to adverse events or intolerability.
* Willing and able to comply with study procedures.
* Able to provide written informed consent.

Exclusion Criteria

* Unwilling or unable to provide written informed consent and to comply with study procedures.
* Any patient for whom providing a buccal swab sample would be contraindicated or not possible.
* Subjects diagnosed as not having anxiety or depression.
* Patients at significant risk for suicide and/or in need of immediate hospitalization as judged by the investigator.
* Diagnosis of Bipolar Disorder, as assessed by patient history or M.I.N.I. response.
* Diagnosis of Schizophrenia or Schizoaffective disorder, as assessed by patient history or M.I.N.I. response.
* History or diagnosis of a personality disorder, as assessed by patient history or M.I.N.I. response.
* History of physical traumatic injury (i.e., TBI) resulting in depression.
* Patients new to psychotherapy (provided by licensed and trained mental health professionals) or have not been on a stable psychotherapy regimen for at least 8 weeks.
* Patients receiving other alternative treatments such as Electroconvulsive Therapy (ECT), Transcranial Magnetic Stimulation (TMS), Vagal Nerve Stimulation (VNS), and Deep Brain Stimulation (DBS).
* Patients with a history of chronic renal dysfunction, Chronic Kidney Disease (Stage 4 or 5).
* Patients with abnormal hepatic function within the last 2 years, (INR >1.2 not attributable to anticoagulant medications, AST/aspartate aminotransferase or ALT/alanine aminotransferase >1.5x normal, or suspected cirrhosis).
* Patients with a history of malabsorption (short gut syndrome).
* Patients with any gastric or small bowel surgery less than 3 months prior to study enrollment.
* Patients with significant unstable medical condition, neurological disorders (e.g. epilepsy, Parkinson's disease or stroke) or life threatening disease.
* Patients who are currently being treated for anxiety and /or depression incorporating pharmacogenetic information.
* History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic for 6 months.
* Patients with any significant substance use disorder as assessed by M.I.N.I. response and judged by the investigator.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The reduction of adverse drug events (ADE) subsequent to pharmacogenetics-guided treatment as compared to standard of care for treatment of depression and/or anxiety symptoms. | 12 weeks

SECONDARY OUTCOMES:
Change in the Hamilton Rating Scale for Depression (HAMD-17) score from baseline. | 12 weeks
Change in the Hamilton Rating Scale for Anxiety (HAM-A) score from baseline. | 12 weeks
Percentage of depression subjects who respond (≥50% decrease in HAM-D17 from baseline or remit, HAM-D17 total score ≤7). | 12 weeks
Percentage of anxiety subjects who respond (≥50% decrease in HAM-A from baseline or remit, HAM-A total score ≤7) | 12 weeks
Time to response/remission of depressive symptoms. | 12 weeks
Time to response/remission of anxiety symptoms. | 12 weeks
Medication change: Number of subjects who changed their antidepressant and anxiety medication regimens from baseline. | 12 weeks
The impact of pharmacogenetic-guided treatment.care costs as measured by HMWDQ | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Centeno, Study Director — AltheaDx
Locations (17):
- United States (17):
  - Adnab Research, Rolling Hills, California
  - Artemis Clinical Research, San Diego, California
  - Adnab Research, Torrance, California
  - Collaborative Neuroscience Network, Torrance, California
  - Innovative Clinical Research, Lauderhill, Florida
  - Innova Clinical Trials, Miami, Florida
  - APG Research, Orlando, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Medpharmics, Metairie, Louisiana
  - Meridian Clinical Research, Norfolk, Nebraska
  - United Medical Associates, Binghamton, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Carolina Partners in Mental HealthCare, Raleigh, North Carolina
  - Detweiler Family Medicine, Lansdale, Pennsylvania
  - Relaro Medical Trials, Dallas, Texas
  - Tidewater Clinical Research, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley P, Shiekh M, Mehra V, Vrbicky K, Layle S, Olson MC, Maciel A, Cullors A, Garces JA, Lukowiak AA. Improved efficacy with targeted pharmacogenetic-guided treatment of patients with depression and anxiety: A randomized clinical trial demonstrating clinical utility. J Psychiatr Res. 2018 Jan;96:100-107. doi: 10.1016/j.jpsychires.2017.09.024. Epub 2017 Sep 23. PMID 28992526